CLINICAL TRIAL: NCT05220436
Title: DISCOVER "Getting the Life You Want" Workshop Programme for Care Experienced Young People Aged 16-19: A Feasibility and Acceptability Pilot Study
Brief Title: DISCOVER Workshop Programme for Care Experienced Young People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: South London and Maudsley NHS Foundation Trust (Other)
Collaborators: Medway Children's Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 303093
Record Dates: First submitted 2021-10-13; First posted 2022-02-02 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Mental Health Issue; Emotional Stress; Emotional Regulation
Keywords: CARE LEAVERS; LOOKED AFTER CHILDREN; PSYCHOLOGICAL INTERVENTION; WORKSHOP PROGRAMME; ADAPTATION; COGNITIVE BEHAVIOUR THERAPY; ACCEPTANCE AND COMMITMENT THERAPY
MeSH Terms: conditions — Stress, Psychological; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DISCOVER workshop programme (Experimental): As this is a case series study, all participants will receive the intervention (i.e. no other arms to the study design).
  The DISCOVER workshop programme includes: 1:1 mental health and emotional well-being assessment session with a Clinical Psychologist, a group workshop day, follow-up supportive phone calls and a closing follow-up 1:1 mental health and emotional well-being session with a Clinical Psychologist.
  Interventions: Other: DISCOVER workshop programme

INTERVENTIONS:
Other: DISCOVER workshop programme — See arm description. The manualised group workshop day is informed by Cognitive Behaviour Therapy and Acceptance & Commitment Therapy principles.
  Other Names: DISCOVER "Getting the Life You Want"

SUMMARY:
The NHS DISCOVER team has secured 2-year funding from the Maudsley Charity to tailor the workshop programme the investigators deliver in school Sixth Forms to meet the specific needs of Care Experienced young people. The investigators are planning to complete a pilot of this adapted workshop programme within Medway Children's Social Services to explore its feasibility, accessibility, acceptability and early-stage efficacy within this population of adolescents.

Investigators from the DISCOVER team will recruit young people aged 16-19yrs who are currently known to the Medway Care Leavers 16+ teams. The study will be conducted at Medway Local Authority sites, with the option of some stages being completed remotely via Microsoft Teams if needed in the context of the ongoing COVID-19 pandemic.

ELIGIBILITY:
Inclusion Criteria:

Participants who are eligible to take part in this DISCOVER research project will be:

* Young people aged 16-19 years who have experience of being in Care and are currently under one of the Medway Children's Social Care, Care Leavers 16+ teams. This means that they are either currently a Looked After young person or a Care Leaver (i.e. they are no longer Looked After but they remain under the care of a Medway Care Leavers team).
* Able to work within a group setting over the course of a day workshop.
* Able to communicate and read in English.

Exclusion Criteria:

The investigators will not be able to recruit young people to the project if they are:

* Acutely psychotic or actively suicidal.
* Currently taking part in other research project(s).
* Under the influence of alcohol or any other substances during DISCOVER programme meetings - this is essential as a safety consideration for all participants and staff. Struggles with alcohol/substance use in themselves are not necessarily grounds for exclusion; the investigators will discuss with the allocated member of the young person's Care Leavers 16+ team on a case-by-case basis where relevant.
* Unable to communicate and read in English - as the investigators are at an early stage in developing this DISCOVER workshop programme for Care Experienced young people, these young people must be excluded at this time. However, the investigators are eager to review this criterion in future to enhance the accessibility of the intervention, once the initial feasibility and acceptability of the workshop programme has been established.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Sclare, DClinPsy, Principal Investigator — NHS DISCOVER Team, South London & Maudsley NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - 16+ Care Leavers Service, Medway Children's Services, Chatham
  - South London & Maudsley NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Our funder - Maudsley Charity - summarise the planned project on their website — https://maudsleycharity.org/case-studies/an-app-to-help-young-people-with-anxiety/

RESULTS

PARTICIPANT FLOW:
Groups:
- DISCOVER Workshop Programme: As this is a case series study, all participants will receive the intervention (i.e. no other arms to the study design).
  The DISCOVER workshop programme includes: 1:1 mental health and emotional well-being assessment session with a Clinical Psychologist, a group workshop day, follow-up supportive phone calls and a closing follow-up 1:1 mental health and emotional well-being session with a Clinical Psychologist.
  DISCOVER workshop programme: See arm description. The manualised group workshop day is informed by Cognitive Behaviour Therapy and Acceptance & Commitment Therapy principles.
Period: Overall Study
Arm/Group | DISCOVER Workshop Programme
Started | 10
Completed | 7
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 10
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.82 (1.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: White British | 8
  Ethnicity: British Asian: Other | 1
  Ethnicity: Other Mixed Background | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 10

OUTCOME MEASURES:

1. Primary Outcome: Participant Uptake (Feasibility & Acceptability)
Description: Number of young people who come forward for and ultimately take part in the new DISCOVER workshop programme
Time Frame: From outset of recruitment, through to final study completion: 7 months
Population: 10 Care Experienced young peopled aged 16-19yrs consented to take part in the DISCOVER GtLYW study.
Measure: Count of Participants; unit: Participants
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 10
Participants | 10

2. Primary Outcome: Participant Retention (Feasibility & Acceptability)
Description: Number of young people who remain in the study throughout all stages of the programme
Time Frame: From outset of recruitment, through to final study completion: 7 months
Population: Seven 16-19yr old Care Experienced young people completed the full workshop programme.
Measure: Count of Participants; unit: Participants
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 10
Participants | 7

3. Primary Outcome: Participant Feedback About Experience of the Programme (Acceptability)
Description: Anonymous workshop feedback survey Semi-structured interview to gather participants' qualitative feedback about the programme
Time Frame: At the end of the workshop day and during closing follow-up one-to-one meeting with DISCOVER team: 2 months later
Population: Young people who attended were asked to provide anonymised feedback at the end of their DISCOVER workshop day. Their qualitative feedback response were gathered during the final 1:1 DISCOVER meeting at the end of the programme.
Measure: Count of Participants; unit: Participants
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 7
Participants
  No. young people who rated the quality of the DISCOVER service on the workshop day as excellent/good | 7
  No. young people who reported that they were satisfied with the DISCOVER service on the workshop day | 7
  No. young people who reported that they felt that they got the help they wanted on the workshop day. | 7
  No. young people who rated that 'all' or 'most' of their needs had been met on the workshop day. | 7
  No. young people reported that they would recommend the workshop to a friend. | 7

4. Secondary Outcome: Mood and Feelings Questionnaire (Angold et al., 1995)
Description: Depression/low mood symptoms (self-report) - Scores range from 0-66 - higher score indicates higher level of depression symptoms
Time Frame: CHANGE MEASURE: Pre-workshop and follow-up one-to-one meetings (Baseline - 2 months after workshop day)
Population: As per description for previous outcomes (the same 7 young people who completed the full DISCOVER GtLYW programme).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 7
score on a scale
  Pre-intervention | 25.57 (9.36)
  Post-intervention | 18.43 (9.68)

5. Secondary Outcome: The Screen for Child Anxiety Related Disorders (Birmaher et al, 1999)
Description: Anxiety symptoms (self-report) - Scores range from 0-82 - higher score indicates higher level of anxiety
Time Frame: CHANGE MEASURE: Pre- and post-workshop 1:1 meetings (Baseline - 2 months after workshop day)
Population: As per description for previous outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 7
score on a scale
  Pre-intervention | 47.71 (10.05)
  Post-intervention | 30.86 (15.60)

6. Secondary Outcome: Child & Adolescent Mindfulness Measure (Greco et al., 2011)
Description: Capacity for mindfulness (self-report) - Scores range from 0-40 - higher score indicates higher level of mindfulness (after reverse scoring)
Time Frame: CHANGE MEASURE: Pre-workshop and follow-up one-to-one meetings (Baseline - 2 months after workshop day)
Population: As per description for previous outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 7
score on a scale
  Pre-intervention | 15.43 (3.69)
  Post-intervention | 23.57 (6.00)

7. Secondary Outcome: Warwick & Edinburgh Mental Well-Being Scale (Tennant et al., 2007)
Description: Emotional well-being and resilience (self-report) - Scores range from 14-70 - higher score indicates greater positive mental wellbeing
Time Frame: CHANGE MEASURE: Pre-workshop and follow-up one-to-one meetings (Baseline - 2 months after workshop day)
Population: As per description for previous outcomes.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DISCOVER Workshop Programme
Number analyzed (Participants) | 7
score on a scale
  Pre-intervention | 41.86 (8.53)
  Post-intervention | 42.56 (6.47)

ADVERSE EVENTS:
Time Frame: The full study lasted between 03/01/2022 - 31/03/2023. Each young person's journey through the study lasted 2-3 months, depending on when they were available for their closing DISCOVER 1:1 meeting at the end of the programme.
Description: We did not use a formal metric of adverse event collection, but rather gathered information about the wellbeing of our participants (young people and staff) throughout regular communication with our project partners within the Medway Care Leavers service.
Arm/Group | DISCOVER Workshop Programme
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/36/NCT05220436/Prot_SAP_000.pdf